CLINICAL TRIAL: NCT05789459
Title: Comparison of Outcomes With Stapler Versus Hand-Sewn Closure of the Pancreatic Stump Following Minimally Invasive Distal Pancreatectomy: A Retrospective Cohort Study
Brief Title: Comparison of Outcomes With Stapler Versus Hand-Sewn Closure After Minimally Invasive Distal Pancreatectomy
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Other Study IDs: DP-POPF
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Distal Pancreatectomy; Postoperative Pancreatic Fistula
MeSH Terms: interventions — Surgical Staplers; Sutures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stapler group: closure with a stapler
  Interventions: Device: Stapler
- Hand-sewn group: closure with suture
  Interventions: Other: Suture

INTERVENTIONS:
Device: Stapler — Stapler
  Groups: Stapler group
Other: Suture — Suture
  Groups: Hand-sewn group

SUMMARY:
The incidence of postoperative pancreatic fistula (POPF) after Distal pancreatectomy (DP) remains high. Of the available mitigation strategies, high-quality closure of the pancreatic stump is fundamental.

Researchers failed to find a decrease in the incidence of POPF after stapler closure of the pancreatic stump compared with that related to hand-sewn suture in DP. Minimally invasive DP (MDP) is becoming the first choice for patients and surgeons, few studies have evaluated whether stapler closure is superior to hand-sewn suture for stump closure in MDP.

Therefore, this retrospective study was aimed at evaluating the effect of stapler versus hand-sewn closure on the incidence of POPF after MDP.

ELIGIBILITY:
Inclusion Criteria:

* Underwent elective minimally invasive pancreatic body and tail resection with or without splenectomy

Exclusion Criteria:

* Incomplete medical records
* History of previous pancreatic operations
* Emergent operation
* Conversion to open pancreatectomy
* Receipt of wedge resection or other procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent MDP in our institution between July 2018 and June 2021.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pancreatic fistula (POPF) | Within 3 months after pancreatic surgery
  The outcome was POPF per the International Study Group of Pancreatic Surgery definition

SECONDARY OUTCOMES:
delayed gastric emptying (DGE) | Within 3 months after pancreatic surgery
  identified and graded according to the ISGPS criteria
postpancreatectomy hemorrhage (PPH) | Within 3 months after pancreatic surgery
  identified and graded according to the ISGPS criteria
Chyle leak | Within 3 months after pancreatic surgery
  identified and graded according to the ISGPS criteria
Surgical complications | Within 3 months after pancreatic surgery
  classified according to the Clavien-Dindo system

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, Principal Investigator — Zhejiang University
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China